CLINICAL TRIAL: NCT06440226
Title: Behaviors Of Boredom, Memory, and Wakefulness, and Their Relation to Determining the Frequency of Lucid Dreaming
Brief Title: Testing Methods to Increase the Frequency of Lucid Dreaming
Acronym: RRF
Status: Completed | Type: Observational
Sponsor: Abdulraheem Mohamed Gouda (Other)
Responsible Party: Sponsor-Investigator, Abdulraheem Mohamed Gouda, Research Director, Reserology Research Foundation
Organization: Reserology Research Foundation (Other)
Other Study IDs: ReserologyRF; Grantee 000010000 (Other: Reserology Research Foundation)
Record Dates: First submitted 2024-05-21; First posted 2024-06-03 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Sleep Wake Disorders
Keywords: sleep; sleep disorder; lucid dreaming; dreams; sleep hygiene
MeSH Terms: conditions — Sleep Wake Disorders; Sleep Hygiene

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — All records of participants and randomly selected individuals are kept.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Placebo Group: Detailed in study, no dosages, no drugs used.
- Actual Group: Detailed in study, no dosages, no drugs used.
  Interventions: Behavioral: Eye Movement Technique; Behavioral: Memory Recall of Previous Night's Thoughts; Behavioral: Recall of Previous Lucid Dreams
- Standard Assessment Group: Detailed in study, no dosages, no drugs used.

INTERVENTIONS:
Behavioral: Eye Movement Technique — Participants were instructed to move their eyes as much as possible with their eyes closed just before falling asleep. This technique aimed to mimic the Rapid Eye Movement (REM) sleep phase, which is often associated with more vivid and memorable dreams.
  Groups: Actual Group
Behavioral: Memory Recall of Previous Night's Thoughts — Another intervention involved asking participants to recall and think about their thoughts or events from the previous night before going to sleep. This method engaged cognitive processes related to memory and reflection, potentially setting the stage for increased awareness during sleep.
  Groups: Actual Group
Behavioral: Recall of Previous Lucid Dreams — Participants were also asked to recall their lucid dreams from previous nights. This intervention seemed to activate memory and awareness related to dreaming, which significantly increased the likelihood of experiencing lucid dreams the following night.
  Groups: Actual Group

SUMMARY:
This study investigates the impact of lucid dreaming on individuals and explores methods to increase the likelihood of inducing lucid dreams intentionally. This study explores the impact of lucid dreaming on individuals, examining how this unique state of consciousness affects mental and emotional well-being. It further explores various methods aimed at increasing the likelihood of intentionally inducing lucid dreams. By analyzing scientific literature and experimental findings, the research highlights the potential therapeutic and creative benefits of lucid dreaming. Additionally, the study offers practical techniques designed to enhance the frequency of lucid dreams, such as maintaining a dream journal, eye movement before sleep, and recall of memories. These approaches provide individuals with tools to harness the power of lucid dreaming for personal growth and self-discovery.This study highlights the potential benefits of lucid dreaming and provides practical techniques for enhancing its frequency.

DETAILED DESCRIPTION:
This detailed study explores the profound impact of lucid dreaming on individuals and assesses various techniques designed to intentionally induce lucid dreams. Lucid dreaming, where dreamers are aware that they are dreaming and can often control their dreams' content, has long intrigued both the scientific community and the general public due to its potential for deep psychological insight and self-improvement.

The primary objective of the research was to investigate methods that could significantly increase the likelihood of inducing lucid dreams.

In continuation, the study explores various methodologies aimed at increasing the probability of individuals intentionally inducing lucid dreams. Techniques such as targeted memory reactivation, where dreamers set intentions before sleep, are scrutinized for their effectiveness. The research examines how these methods align with neuroscientific understandings of sleep phases, particularly REM sleep when lucid dreaming most frequently occurs. The correlation between sleep quality, dream recall frequency, and the propensity to experience lucid dreams is highlighted, proposing that enhancing one's sleep hygiene could indirectly foster the conditions suitable for lucid dreaming.

Analyzing extensive scientific literature and experimental data, the study discusses the uses of lucid dreaming as a cognitive tool. It examines scenarios that promote problem-solving and creative thinking through conscious navigation and manipulation of dream content. This allows individuals to rehearse skills, resolve conflicts, and explore creative avenues that may not be accessible in waking life.

Lastly, these approaches offer individuals practical tools to harness the power of lucid dreaming for personal growth and self-discovery. The study emphasizes the importance of intentionality in entering the lucid dreaming state and maintaining a mindset conducive to this during waking hours. The capacity to engage in lucid dreaming is presented as a meaningful pursuit that can contribute to one's mental health and creative expression, fostering a deeper understanding and appreciation of this complex cognitive phenomenon.

ELIGIBILITY:
Inclusion Criteria:

* Normal blood pressure, Healthy weight, no record of sleep apnea, no difficulty sleeping, ages between 18-30 only.

Exclusion Criteria:

* Overweight(muscle being taken into consideration, not using BMI), high or low blood pressure,

Ages: 18 Years to 30 Years | Sex: All
Age Groups: Adult
Study Population: Young, healthy, individuals with no previous record of medical sleep conditions.
Sampling Method: Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2024-01-09 (Actual); Primary Completion 2024-04-26 (Actual); Study Completion 2024-05-02 (Actual)

PRIMARY OUTCOMES:
Testing the likelihood of Lucid Dreaming in Participants | 4 months
  Measuring the likelihood of lucid dreaming with the implementation of the methods mentioned in the behavioural section of this study.

CONTACTS AND LOCATIONS:
Overall Officials: Abdelraheem Mohamed, Study Chair — Reserology Research Foundation
Locations (1):
- Reserology Research, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Privacy reasons as requested by participants when signed up contractually.

REFERENCES:
- [Result] Greenwald B, Lombard LA, Watanabe TK. Managing sleepiness after traumatic brain injury. PM R. 2011 May;3(5):480-5. doi: 10.1016/j.pmrj.2011.04.010. No abstract available. PMID 21570037